CLINICAL TRIAL: NCT00484003
Title: A 3-Month Open Label, National, Quality of Life , and Safety Study With Pimecrolimus Cream, 1% in Children (Age 2-12 Years ) With Atopic Dermatitis
Brief Title: A Quality of Life and Safety Study With Pimecrolimus Cream, 1% in Children (Age 2-12 Years) With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASM981CZA01
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Atopic Eczema
Keywords: Atopic eczema; Pimecrolimus; Children; Quality of life; Safety; Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus cream 1%
  Other Names: Elidel

SUMMARY:
The study will evaluate the safety and effect of pimecrolimus cream 1% on quality of life of caregivers of South African children with mild to moderate atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥2 years ≤12 years of age
* Atopic dermatitis on sensitive skin areas only ( i.e. face , neck and flexures )
* Subjects in whom other treatment modalities are inadvisable according to the investigator's clinical opinion or have failed on other treatment modalities due to intolerance or inadequate response.
* Patients with a history of mild to moderate AD
* Subjects should present at visit 1 with a clear clinical diagnosis of mild to moderate AD.
* Subject's parents or legal guardian must have been informed of the study procedures and must have signed the Informed Consent form approved for the study prior to any study related procedures

Exclusion Criteria:

* Subjects who have active viral infections at the site(s) of treatment. In the presence of other dermatological infections, the use of appropriate antimicrobial agents should be instituted.
* Subjects who present with systemic malignancy or active lymphoproliferative diseases/disorders (e.g., lymphoma, neoplastic disease, chronic lymphoproliferation).
* Subjects who present with clinical conditions other than AD that can, in the opinion of the investigator, interfere with the evaluation
* Subjects who are receiving photo-therapy (e.g., PUVA, UVB) or immunosuppressive therapy (e.g., cyclosporine, FK-506 [tacrolimus]).
* Subjects who have used investigational drugs within 8 weeks prior to first application of study medication or intended use of other investigational drugs during the course of this study.
* Subjects who have used, or are using 0.03% or 0.1% tacrolimus ointment.
* Pimecrolimus cream 1% is contraindicated in subjects who have known or suspected hypersensitivity to pimecrolimus or any components of the cream
* Subjects not medically stable or subjects with any condition which, in the opinion of the investigator, should render the subject ineligible for the study.
* Pregnancy and lactation (if applicable)
* Pimecrolimus cream 1% should not be used during pregnancy or lactation

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-10; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life assessment on scheduled visits at Day 1 (Baseline), Day 14 and Day 90 or day of early discontinuation visit.

SECONDARY OUTCOMES:
Safety data will be collected by monitoring and recording all adverse events (AEs)and Serious Adverse Events(SAEs) throughout the duration of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative Sites, Various Cities, South Africa